CLINICAL TRIAL: NCT01388894
Title: Functional MRI and MRA in Migraine With Aura
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Jes Olesen, Danish Headache Center
Other Study IDs: MA-01
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-05

CONDITIONS: Migraine With Aura
MeSH Terms: conditions — Migraine with Aura

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients who report that exposure to bright light or strenuous physical activity will induce migraine aura will be provoked using one or both of these methods. Followingly the patients will be examined by functional MRI. Íf the patients develop migraine headache, MR angiography will be performed as well. The primary study hypothesis is that the functional MRI signal will show features similar to those of the electrophysiological phenomenon of cortical spreading depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with migraine with aura as defined by The International Classification of Headache Disorders 2
* Age between 18 and 80 years both inclusive
* Reports that bright light or strenuous physical activity may trigger migraine aura

Exclusion Criteria:

* Contraindications towards exposure to photostimulation or strenuous exercise
* Body weight above 130 kg
* Pregnant or lactating females
* Contraindications towards MRI scanning
* History or clinical signs of: cardiovascular disease, psychiatric disease, substance abuse or any symptom or disease considered relevant by the examining physician.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with migraine with aura
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-12

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark